CLINICAL TRIAL: NCT00450177
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial of the Effects of Enteral Iron Supplementation on Anemia and Risk of Infection in Critical Illness
Brief Title: Efficacy of Enteral Iron Supplementation in Critical Illness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 052007738
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Anemic, Critically Ill Patients
Keywords: iron; critical illness; anemia; infection
MeSH Terms: conditions — Critical Illness; Anemia; Infections | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron Group (Experimental): Ferrous sulfate 325 mg either by capsule or oral solution three times a day at 9 am, 1pm and 5 pm until hospital discharge or for 42 days, whichever occurs first.
  Interventions: Drug: Ferrous Sulfate
- Placebo Group (Placebo Comparator): Placebo capsule three times a day at 9 am, 1pm and 5 pm until hospital discharge or for 42 days, whichever occurs first.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Ferrous Sulfate — Iron group
  Arms: Iron Group
Drug: Placebo Oral Tablet — Placebo group
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to investigate the efficacy of enteral iron supplementation for improving anemia, decreasing the risk of blood transfusion, and decreasing mortality in patients who are hospitalized in the intensive care unit. This study will also address any relationship between enteral iron supplementation and risk of infection.

DETAILED DESCRIPTION:
Critical illness is characterized by the anemia of inflammation, which is partially caused by sequestration of iron from bone marrow sites of erythropoiesis into storage within the reticuloendothelial system as ferritin. Also the majority of critically ill patients are hypoferremia, the efficacy of iron supplementation remains unknown. Furthermore, several retrospective studies have found an association between iron overload and infection. However, the relative risk/benefit profile of enteral iron supplementation with respect to infection has not been studied. The purpose of this study is to evaluate the efficacy of enteral iron supplementation in critically ill patients. The hypothesis is that enteral iron supplementation will result in both an improved hematocrit and a decreased need for blood transfusion, without increasing the risk of infection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Anemia (Hemoglobin < 13.0 g/dL)
* ≤ 72 hours from hospital admission
* Current tolerance of enteral medications
* Expected ICU LOS > 5 days

Exclusion Criteria:

* Active bleeding
* Chronic inflammatory disease
* End-stage renal disease
* Hematologic disorders
* Macrocytic anemia
* Current use of erythropoietin
* Pregnancy
* Prohibition of RBC transfusions
* Moribund state in which death is imminent
* Enrollment in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip S Barie, MD, MBA, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Derived] Pieracci FM, Henderson P, Rodney JR, Holena DN, Genisca A, Ip I, Benkert S, Hydo LJ, Eachempati SR, Shou J, Barie PS. Randomized, double-blind, placebo-controlled trial of effects of enteral iron supplementation on anemia and risk of infection during surgical critical illness. Surg Infect (Larchmt). 2009 Feb;10(1):9-19. doi: 10.1089/sur.2008.043. PMID 19245362

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iron Group | Placebo Group
Started | 97 | 103
Completed | 88 | 92
Not Completed | 9 | 11
Not completed — Adverse Event | 7 | 4
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Withdrawal by Primary Team | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Group | Placebo Group | Total
Number analyzed (Participants) | 97 | 103 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (1.9) | 58.2 (1.7) | 57.0 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 55 | 103
  Male | 49 | 48 | 97
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline hematocrit [Mean (Standard Deviation); unit: % of RBC in total blood volume] | 32.0 (0.5) | 31.9 (0.4) | 31.9 (0.4)
Baseline MCV [Mean (Standard Deviation); unit: femtoliters] — Mean Corpuscular Volume (MCV)
  femtoliters | 88.7 (0.7) | 88.6 (0.8) | 88.6 (0.8)
Baseline EBL [Mean (Standard Deviation); unit: milliliters] — Estimated Blood Loss (EBL)
  milliliters | 171 (45) | 207 (50) | 189 (48)
Baseline RBC transfusion [Count of Participants; unit: Participants] — Red Blood Cell (RBC)
  Participants | 9 | 19 | 28
Baseline RBC transfusion [Mean (Standard Deviation); unit: milliliters] — Red Blood Cell (RBC)
  milliliters | 135 (58) | 303 (110) | 222 (85)
Admission to enrollment [Mean (Standard Deviation); unit: days] | 1.6 (0.1) | 1.7 (0.1) | 1.7 (0.1)
Admission APACHE II [Mean (Standard Deviation); unit: units on a scale] — Acute Physiology and Chronic Health Evaluation (APACHE): Designed to measure the severity of disease for adult patients admitted to intensive care units. The point score is calculated from a patient's age and 12 routine physiological measurements: alveolar-arterial oxygen gradient or arterial blood gasses, temperature, mean arterial pressure, pH arterial, heart rate, respiratory rate, sodium (serum), potassium (serum), creatinine, hematocrit, white blood cell count, glasgow coma scale. The APACHE score ranges from 0 to 71, with 0 indicating a higher mortality risk and 71 a lower risk.
  units on a scale | 15.9 (0.8) | 14.9 (0.8) | 15.4 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Hematocrit
Time Frame: Day 7, Day 14, Day 21, Day 28
Measure: Mean (Standard Deviation); unit: percentage of RBC in blood
Arm/Group | Iron Group | Placebo Group
Number analyzed (Participants) | 97 | 103
percentage of RBC in blood
  Day 7 | 29.3 (0.5) | 29.1 (0.5)
  Day 14 | 28.6 (0.4) | 28.2 (0.5)
  Day 21 | 29.2 (0.4) | 28.1 (0.6)
  Day 28 | 27.8 (0.6) | 28.1 (0.5)

2. Primary Outcome: Serum Iron Concentration
Time Frame: Day 7, Day 14, Day 21, Day 28
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Iron Group | Placebo Group
Number analyzed (Participants) | 97 | 103
mcg/mL
  Day 7 | 35 (0.6) | 37 (0.7)
  Day 14 | 34 (0.5) | 34 (0.7)
  Day 21 | 34 (0.6) | 40 (0.6)
  Day 28 | 37 (0.5) | 36 (0.7)

3. Primary Outcome: Serum Ferritin Concentration
Time Frame: Day 7, Day 14, Day 21, Day 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iron Group | Placebo Group
Number analyzed (Participants) | 97 | 103
ng/mL
  Day 7 | 280 (46) | 265 (73)
  Day 14 | 268 (51) | 268 (80)
  Day 21 | 251 (40) | 355 (83)
  Day 28 | 383 (54) | 361 (76)

4. Primary Outcome: Erythrocyte Zinc Protoporphyrin Concentration
Time Frame: Day 7, Day 14, Day 21, Day 28
Measure: Mean (Standard Deviation); unit: micromol:mol heme
Arm/Group | Iron Group | Placebo Group
Number analyzed (Participants) | 97 | 103
micromol:mol heme
  Day 7 | 69 (4) | 67 (5)
  Day 14 | 75 (6) | 77 (5)
  Day 21 | 86 (5) | 91 (6)
  Day 28 | 84 (6) | 89 (5)

5. Secondary Outcome: Number of Subjects That Received at Least One RBC Transfusion During Admission to the Hospital
Time Frame: Throughout hospital stay up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Group | Placebo Group
Number analyzed (Participants) | 97 | 103
Participants | 29 | 46
Statistical Analysis 1: Comparison: Iron Group vs Placebo Group; Test type: Other; p = 0.03, Chi-squared

6. Secondary Outcome: Number of Subjects That Incurred at Least One Infection Throughout Hospital Admission
Time Frame: Throughout hospital stay up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Group | Placebo Group
Number analyzed (Participants) | 97 | 103
Participants | 45 | 48

7. Secondary Outcome: Instance of Drug-related Constipation Throughout Hospital Admission
Time Frame: Throughout hospital stay up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Group | Placebo Group
Number analyzed (Participants) | 97 | 103
Participants | 12 | 9

8. Secondary Outcome: Average Number of Days That Subjects Were Taking Antibiotics
Time Frame: Throughout hospital stay up to 6 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Iron Group | Placebo Group
Number analyzed (Participants) | 97 | 103
days | 14 (2) | 16 (3)

9. Secondary Outcome: Hospital Mortality, as Measured by Number of Subject Deaths While Admitted to Hospital
Time Frame: Throughout hospital stay up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Group | Placebo Group
Number analyzed (Participants) | 97 | 103
Participants | 9 | 10

10. Secondary Outcome: Average Length of Stay in the Hospital
Time Frame: Throughout hospital stay up to 6 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Iron Group | Placebo Group
Number analyzed (Participants) | 97 | 103
days | 14 (1) | 16 (2)

ADVERSE EVENTS:
Arm/Group | Iron Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/103
Other Adverse Events (participants affected / at risk) | 7/97 | 4/103
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iron Group (N=97) | Placebo Group (N=103)
Gastrointestinal upset (Gastrointestinal disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No